CLINICAL TRIAL: NCT04399980
Title: Mavrilimumab to Reduce Progression of Acute Respiratory Failure in Patients With Severe COVID-19 Pneumonia and Systemic Hyper-inflammation
Brief Title: Mavrilimumab to Reduce Progression of Acute Respiratory Failure in COVID-19 Pneumonia and Systemic Hyper-inflammation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Kiniksa Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IND 149324; IRB 20-523 (Other: Cleveland Clinic IRB)
Record Dates: First submitted 2020-05-21; First posted 2020-05-22 (Actual); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: COVID 19; SARS-CoV 2; Pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — mavrilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Treatment infusion
  Interventions: Drug: Mavrilimumab
- Control (Placebo Comparator): Placebo infusion
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Mavrilimumab — Treatment infusion
  Other Names: KPL-301
  Arms: Intervention
Drug: Placebos — Placebo infusion
  Other Names: Control
  Arms: Control

SUMMARY:
The purpose of this prospective, Phase 2, multicenter, blinded, randomized placebo controlled study is to demonstrate that early treatment with mavrilimumab prevents progression of respiratory failure in patients with severe COVID-19 pneumonia and clinical and biological features of hyper-inflammation.

DETAILED DESCRIPTION:
This prospective, Phase 2, multi-center, blinded randomized placebo-controlled study is designed to demonstrate that early treatment with mavrilimumab prevents progression of respiratory failure in patients with severe Covid-19 pneumonia and clinical and biological features of hyper-inflammation.

The study population includes patients who have severe pneumonia, defined as hospitalization due to Covid-19 with abnormal chest imaging and SpO2 <92% on room air or requirement for supplemental oxygen.

Enrollment: The study will be performed in approximately 4 months total, starting from the first patient enrolled with enrollment expected to complete within 2 months.

Follow-up period: The follow-up period is 60 days for each patient enrolled.

A total of 60 patients will be randomized using a 1:1 allocation ratio: 30 subjects will receive mavrilimumab, and 30 subjects will receive placebo infusion. The investigator, clinical team, and subject will be blinded to treatment assignment.

Participants will be identified by regular review of hospitalized COVID19 patients to evaluate for inclusion and exclusion criteria. Participants will then be approached in the standard manner by study investigator and coordinator/research nurse.

Research interventions will take place in the hospital in accordance with privacy standards.

The study team is informed on all study procedures and requirements with daily meetings and the opportunity to continuously update through secure channels.

In this multicenter consortium, each participating site will have their own IND for patients enrolled at their site. Data collection will occur at each of the 4 academic centers, and data analysis and randomization scheme will be performed by one site, Cleveland Clinic C5 Research.

ELIGIBILITY:
Inclusion Criteria (must meet all):

1. Written informed consent must be obtained before any assessment is performed
2. Documented COVID19 pneumonia defined as positive SARS-CoV2 test AND abnormalities/ infiltrates on chest x-ray or computed tomography AND active fever or documented fever within 24-48 hours or ongoing anti-pyretic use to suppress fever
3. Hypoxia (Room air SpO2 <92% or requirement for supplemental oxygen)
4. Increased serum inflammatory marker (CRP > 5 mg/dL)
5. Severity of disease warrants inpatient hospitalization

Exclusion Criteria:

1. Onset of COVID-19 symptoms >14 days
2. Age < 18 years-old
3. Hospitalized >7 days
4. Mechanically ventilated
5. Serious concomitant illness which in the opinion of the investigator precludes the patient from enrolling in the trial, including (but not limited to):

   * History of immunodeficiency (congenital or acquired)
   * Neutropenia (absolute neutrophil count <1,500/mm3)
   * History of solid-organ or bone marrow transplant
   * History of current systemic autoimmune or autoinflammatory disease(s) requiring systemic immune-modulating drugs
   * History of myeloproliferative disorder or active malignancy receiving cytotoxic chemotherapy
   * Pre-existing severe pulmonary disease (i.e. steroid dependent asthma, COPD on home oxygen, or other restrictive/obstructive lung disease requiring home oxygen)
   * Pre-existing severe left ventricular systolic dysfunction (i.e. LVEF <35%)
   * Known or suspected active tuberculosis (TB), latent TB, or history of incompletely treated TB or at high risk for latent TB (from exposure or prior incarceration)
   * History of active or latent viral hepatitis (i.e. Hepatitis B or C)
   * Concomitant uncontrolled systemic bacterial or fungal infection
   * Concomitant viral infection other than COVID-19 (e.g. Influenza, other respiratory viruses)
   * History of chronic liver disease with portal hypertension
   * History of end-stage renal disease on chronic renal replacement therapy
6. Recent treatment with cell-depleting biological therapies (e.g., anti-CD20) within 12 months, cell-depleting biological therapies (such as anti-tumor necrosis factor [TNF], anakinra, anti-Interleukin [IL]-6 receptor [e.g. tocilizumab], or abatacept) within 8 weeks (or 5 half-lives, whichever is longer), treatment with alkylating agents within 12 weeks, treatment with cyclosporine A, azathioprine, cyclophosphamide, or mycophenolate mofetil (MMF) within 4 weeks
7. Recent treatment with intramuscular live (attenuated) vaccine within 4 weeks
8. Chronic or recent corticosteroid use > 10 mg/day
9. Pregnant. Breast-feeding women are eligible with the decision to continue or discontinue breast-feeding during therapy taking into account the risk of infant exposure, the benefits of breast-feeding to the infant, and benefits of treatment to the mother
10. Enrolled in another investigational study using immunosuppressive therapy
11. Known hypersensitivity to mavrilimumab or any of its excipients
12. In the opinion of the investigator, unable to comply with the requirements to participate in the study
13. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing of investigational drug. Such methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or bilateral tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject
    * Use of oral, (estrogen and progesterone), injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul C Cremer, M. D., Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Cleveland Clinic Florida, Weston, Florida
  - Cleveland Clinic Health System, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cremer PC, Abbate A, Hudock K, McWilliams C, Mehta J, Chang SY, Sheng CC, Van Tassell B, Bonaventura A, Vecchie A, Carey B, Wang Q, Wolski KE, Rajendram P, Duggal A, Wang TS, Paolini JF, Trapnell BC; MASH-COVID study group. Mavrilimumab in patients with severe COVID-19 pneumonia and systemic hyperinflammation (MASH-COVID): an investigator initiated, multicentre, double-blind, randomised, placebo-controlled trial. Lancet Rheumatol. 2021 Jun;3(6):e410-e418. doi: 10.1016/S2665-9913(21)00070-9. Epub 2021 Mar 17. PMID 33754144

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: One-time Mavrilimumab infusion at 6mg/kg via IV
- Control: One-time placebo infusion via IV
Period: Overall Study
Arm/Group | Intervention | Control
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (13.49) | 54.8 (18.44) | 55.75 (15.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 14 | 12 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 8 | 16
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 19 | 40
History of Diabetes [Count of Participants; unit: Participants] | 8 | 9 | 17
History of Hypertension [Count of Participants; unit: Participants] | 10 | 12 | 22
History of Hyperlipidemia [Count of Participants; unit: Participants] | 7 | 11 | 18

OUTCOME MEASURES:

1. Primary Outcome: Subjects Alive and Off of Oxygen at Day 14
Description: Number and percentage of subjects alive and off of oxygen at day 14
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 21 | 19
Participants | 12 | 9

2. Secondary Outcome: Number of Subjects Alive and Without Respiratory Failure at Day 28
Description: Number and percentage of subjects that are alive and without respiratory failure at Day 28
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 21 | 19
Participants | 20 | 15

3. Secondary Outcome: Mortality at Day 28
Description: Number and percentage of patients that expired by Day 28
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 21 | 19
Participants | 1 | 3

ADVERSE EVENTS:
Time Frame: 60 days
Groups:
- Intervention: One-time Mavrilimumab infusion at 6kg/mg via IV
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 1/21 | 4/19
Serious Adverse Events (participants affected / at risk) | 5/21 | 4/19
Other Adverse Events (participants affected / at risk) | 12/21 | 8/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=21) | Control (N=19)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Nausea (General disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Shock (General disorders) | 1 (1) | 0 (0)
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Elevated WBC (Investigations) | 0 (0) | 1 (1)
Hypoxia - Worsening (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=21) | Control (N=19)
Acute Kidney Injury (Renal and urinary disorders) | 4 (4) | 3 (3)
anemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Headache (General disorders) | 0 (0) | 1 (1)
Liver Dysfunction (Hepatobiliary disorders) | 3 (3) | 0 (0)
Shock (General disorders) | 2 (2) | 1 (1)
Pulmonary Embolism (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Investigations) | 1 (1) | 0 (0)
Clot (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Elevated Ferritin (Investigations) | 0 (0) | 1 (1)
Elevated CRP (Investigations) | 0 (0) | 1 (1)
Delirium (Nervous system disorders) | 1 (1) | 1 (1)
Worsening D Dimer (Hepatobiliary disorders) | 0 (0) | 1 (1)
Fever (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Acute Respiratory Syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT04399980/Prot_SAP_001.pdf